CLINICAL TRIAL: NCT05445258
Title: Evaluation of the Safety and Tolerance of the Use of InnoCath AB® Hyper-compliant Balloon Catheters in Peripheral Arteries
Brief Title: Safety and Tolerance of the Use of InnoCath AB® Hyper-compliant Balloon
Acronym: HYPER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Design of the study device will be modified
Sponsor: InnoRa GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: InnoCathAB®_01
Record Dates: First submitted 2022-06-29; First posted 2022-07-06 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Lesions in the Superficial Femoral Artery and/or Popliteal Artery Pars I/II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- InnoCath AB® Balloon (Experimental): endovascular treatment of lesions in the superficial femoral artery (SFA) and/or popliteal artery pars I/II without further luminal widening, and/or for short-term interruption of blood flow with the InnoCath AB® hyper-compliant balloon cathe-ters (100 or 200 mm length)
  Interventions: Device: InnoCath AB® hyper-compliant balloon catheter

INTERVENTIONS:
Device: InnoCath AB® hyper-compliant balloon catheter — endovascular treatment of lesions in the superficial femoral artery (SFA) and/or popliteal artery pars I/II without further luminal widening, and/or for short-term interruption of blood flow with the InnoCath AB® hyper-compliant balloon cathe-ters (100 or 200 mm length)

SUMMARY:
This is a 'first in man' study to demonstrate compliance with the general safety and performance requirements of Regulation (EU) 2017/745 on medical devices (MDR) Annex I as part of the clinical evaluation and for the application of CE-marking. The aim of the study is to evaluate the safety and tolerability of the application and the success rate of the InnoCath AB® hyper-compliant balloon catheter after PTA in peripheral arteries.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Patients with peripheral arterial occlusive disease and intended for endovascular therapy in the SFA and/or popliteal artery pars I/II
* Patients suitable for endovascular therapy in the SFA and/or popliteal artery pars I/II with a hyper-compliant balloon without further luminal widening
* Target vessels with a sufficient "runoff" to the foot with at least one vessel
* Rutherford classification 1-4 if physical and medicinal therapies have not been successful

Exclusion Criteria:

* Aneurysms at the site of inflation
* Application directly in the area of large vessel wall injuries with heavy bleeding
* Rutherford classification 5 and 6

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerance | up to 30 days after intervention
  Number of events, which are related to the medical device being tested

SECONDARY OUTCOMES:
Procedural success | till the end of the procedure
  defined as technical success (ability of the InnoCath AB® hyper-compliant bal-loon catheter to perform as intended, inflation of the device at the lesion site and retraction of the balloon catheter through the introductory sheath) in the ab-sence of vessel rupture, distal embolization, thrombosis, access complications, and major adverse cardiovascular events (cardiac death, myocardial infarction, stroke) as a consequence of the procedure and related to the study device till the end of the procedure
Handling of the InnoCath AB® hyper-compliant balloon catheter | throughout the entirety of the procedure
  The handling of the InnoCath AB® hyper-compliant balloon catheter will be evaluated by the investigator, who assesses various parameters using a scale from 0-2, where 0 describes the better outcome; e.g. balloon deflation and withdrawal of balloon catheter: 0=easy, without any problems, 1=difficult, abnormal, 2=not possible.
Device deficiencies of the InnoCath AB® hyper-compliant balloon catheter | throughout the entirety of the procedure
  The device deficiencies of the InnoCath AB® hyper-compliant balloon catheter will be assessed by the investigator as free-text. Device deficiencies means any inadequacy in the identity, quali-ty, durability, reliability, safety or performance of an investigational device, including malfunc-tion, use errors or inadequacy in information supplied by the manufacturer

CONTACTS AND LOCATIONS:
Overall Officials: Michael Werk, Dr, Principal Investigator — Martin-Luther-Krankenhaus
Locations (2):
- Germany (2):
  - Klinik für Diagnostische und Interventionelle Radiologie Evangelisches Krankenhaus Hubertus, Berlin
  - Klinik für Radiologie und Nuklearmedizin Martin-Luther-Krankenhaus, Berlin

IPD SHARING:
Plan to Share IPD: Undecided